CLINICAL TRIAL: NCT06590740
Title: Establishment of a FeNO Cutoff Value for Evaluating the Response to Budesonide-formoterol in Patients With Chronic Cough Suggestive of Cough Variant Asthma: a Multicenter Prospective Clinical Study
Brief Title: Establish FeNO Cut-off Value for Predicting Budesonide-formoterol Response in Chronic Cough Suggestive of CVA Patients.
Acronym: EFFICIENCY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D589BL00076
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Cough-Variant Asthma
MeSH Terms: conditions — Cough-Variant Asthma | interventions — Budesonide; Formoterol Fumarate; Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Budesonide-Formoterol treatment (Experimental): Budesonide 160 μg/formoterol 4.5 μg, 1 inhalation, BID
  Interventions: Drug: Budesonide-Formoterol treatment

INTERVENTIONS:
Drug: Budesonide-Formoterol treatment — Budesonide 160 μg/formoterol 4.5 μg, 1 inhalation, BID
  Other Names: Budesonide 160 μg/formoterol 4.5 μg treatment

SUMMARY:
This is a multicenter, prospective, single-arm, interventional clinical study to predict the response to budesonide-formoterol treatment in patients with chronic dry or nocturnal cough by determining a cut off value of FeNO. In this study, the response to ICS/LABA treatment is defined as reduction in cough VAS score from baseline of ≥30 mm after 8 weeks of ICS/LABA treatment. Subjects will be treated with Symbicort® 160/4.5 mcg, 1 puff, BID for 8 weeks with 4 study visits: Visit 1 (Day 0), Visit 2 (week 4) and Visit 3, end of study (week 8) and Visit 4, 4 weeks after treatment discontinuation, (week 12). Baseline data will be collected at Day-5 to Day0.

This study will be conducted at around 40 study sites in China. Approximately 1000 patients (age ≥18 years old) with dry cough or nocturnal cough symptoms for at least 8 weeks and no other obvious cause for their cough will be enrolled into this study.

DETAILED DESCRIPTION:
This is a multicenter, prospective, single-arm, interventional clinical study to predict the response to budesonide-formoterol treatment in patients with chronic dry or nocturnal cough by determining a cut off value of FeNO. In this study, the response to ICS/LABA treatment is defined as reduction in cough VAS score from baseline of ≥30 mm after 8 weeks of ICS/LABA treatment. Subjects will be treated with Symbicort® 160/4.5 mcg, 1 puff, BID for 8 weeks with 4 study visits: Visit 1 (Day 0), Visit 2 (week 4) and Visit 3, end of study (week 8) and Visit 4, 4 weeks after treatment discontinuation, (week 12). Baseline data will be collected at Day-5 to Day0.

This study will be conducted at around 40 study sites in China. Approximately 1000 patients (age ≥18 years old) with dry cough or nocturnal cough symptoms for at least 8 weeks and no other obvious cause for their cough will be enrolled into this study. Disclosure Statement: This is an Interventional study with single arm.

Number of Participants:

Approximately 1150 participants will be screened to achieve 1000, based on assuming a screen failure rate of approximately 15%. assigned to study intervention. Study Arms and Duration: Single-arm, 2 months Data Monitoring / Other Committee: Not applicable Statistical Methods： In general, descriptive statistics will be provided for the data collected. For continuous variables, mean, standard deviation, median, quartiles, minimum and maximum will be provided, and for categorical variables, frequency counts and percentages for each category will be provided. Missing data will not be imputed unless otherwise specified. The diagnostic value of FeNO to Budesonide-formoterol response will be measured as the area under the curve (AUC) of the receiver-operating characteristic derived from the Logistic regression model. The study is mainly to investigate if FeNO alone can help to distinguish patients with Budesonide-formoterol response or not, and therefore baseline FeNO value will be the only independent variable included in the model. The optimal cutoff value will be selected by consulting clinical experts, and based on comprehensive assessment of AUC, sensitivity, specificity, PPV, and NPV of different FeNO cut points. To perform discovery and validation within the same study, the total sample will be split randomly into discovery and validation datasets by 70% and 30% respectively. For the validation, similar parameters of diagnostic values will be calculated and compared with those based on the discovery dataset.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily participate in the study and comply with the study requirements, understand, comply with and cooperate with the corresponding examinations, comply with the follow-up schedule, and voluntarily sign the written informed consent form.
2. Patients aged ≥ 18 years.
3. Subjects with cough as the predominant or sole symptom, and manifested as dry or nocturnal cough lasting for ≥ 8 weeks.
4. FEV1/FVC ≥ 70% within 4 weeks from the enrolment.
5. No clinically significant abnormality in the chest CT within 3 months from the enrolment.
6. Cough VAS score ≥ 40 mm measured within 48 hours before enrollment.

Exclusion Criteria:

1. Any history of respiratory infection within 8 weeks from the enrolment.
2. Dyspnea caused by respiratory system disorders.
3. Patients with GERC, upper airway cough syndrome/postnasal drip syndrome as the likely cause of cough.
4. Patients with suspected AECI induced cough.
5. Intolerance to β2 agonists.
6. Used ICS-containing drugs within 8 weeks before enrollment, including ICS or ICS/LABA and so on.
7. Used oral corticosteroids within 8 weeks before enrollment.
8. Used LTRA within 8 weeks before enrollment.
9. Current smokers, or former smokers with a smoking cessation interval of less than 6 months; Smokers with a pack history of greater than 20 pack-years.
10. Individuals with severe respiratory or other systemic diseases.
11. Pregnancy, breast-feeding or planned pregnancy during the study. Fertile women not using acceptable contraceptive measures, as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
To obtain a cut-off value for FeNO which can be used to distinguish responsiveness to 8 weeks treatment of Budesonideformoterol (based on visual analog scale [VAS]). | 8 weeks
  Area under the ROC Curve (AUC), sensitivity, specificity, PPV, NPV

SECONDARY OUTCOMES:
To obtain a cut-off value for FeNO which can be used to distinguish responsiveness to 8 weeks treatment of Budesonideformoterol (based on leicester cough questionnaire [LCQ]). | 8 weeks
  Area under the ROC Curve (AUC), sensitivity, specificity, PPV, NPV
To obtain a cut-off value for FeNO which can be used to distinguish responsiveness to 8 weeks treatment of Budesonideformoterol (based on cough evaluation test [CET]). | 8 weeks
  Area under the ROC Curve (AUC), sensitivity, specificity, PPV, NPV
To assess if the 8 weeks treatment of Budesonide-formoterol response rate differ between the high FeNO group and low FeNO group using the identified cut-off value | 8 weeks
  The response rate in the high FeNO group (those equal or above the new selected FeNO cut point) and the low FeNO group (those below the selected FeNO new cut point).

OTHER OUTCOMES:
To describe patient's characteristic (FeNO) with 8 weeks treatment of Budesonide-formoterol response and those without Budesonideformoterol response. | 8 weeks
  Patient's characteristic: FeNO
To describe patient's characteristic (blood EOS) with 8 weeks treatment of Budesonide-formoterol response and those without Budesonideformoterol response. | 8 weeks
  Patient's characteristic: blood EOS
To describe patient's characteristic (Induced Sputum EOS) with 8 weeks treatment of Budesonide-formoterol response and those without Budesonideformoterol response. | 8 weeks
  Patient's characteristic: Induced Sputum EOS
To describe patient's characteristic (IgE) with 8 weeks treatment of Budesonide-formoterol response and those without Budesonideformoterol response. | 8 weeks
  Patient's characteristic: IgE
To describe patient's characteristic (visual analog scale [VAS]) with 8 weeks treatment of Budesonide-formoterol response and those without Budesonideformoterol response. | 8 weeks
  Patient's characteristic: visual analog scale [VAS]
To describe patient's characteristic (leicester cough questionnaire [LCQ]) with 8 weeks treatment of Budesonide-formoterol response and those without Budesonideformoterol response. | 8 weeks
  Patient's characteristic: leicester cough questionnaire [LCQ]
To describe patient's characteristic (cough evaluation test [CET]) with 8 weeks treatment of Budesonide-formoterol response and those without Budesonideformoterol response. | 8 weeks
  Patient's characteristic: cough evaluation test [CET]
To assess the diagnostic value of EOS in distinguishing responsiveness to 8 weeks treatment of Budesonide-formoterol and determine the optional cutoff value for EOS. | 8 weeks
  AUC, sensitivity, specificity, PPV, NPV
To describe response rate of Budesonideformoterol at 4 and 8 weeks. | 4 weeks, 8 weeks
  Response rate
To explore the bronchial provocation test negative conversion rate in patients with positive baseline provocation test who were treated with budesonide-formoterol for 8 weeks. | 8 weeks
  Bronchial provocation test negative conversion rate.

CONTACTS AND LOCATIONS:
Overall Officials: Kefang Lai, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (32):
- China (32):
  - Research Site, Beijing
  - Research Site, Benxi
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dongguan
  - Research Site, Fenyang
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Heifei
  - Research Site, Heze
  - Research Site, Huizhou
  - Research Site, Jiaxing
  - Research Site, Jinhua
  - Research Site, Liuchow
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanyang
  - Research Site, Quanzhou
  - Research Site, Shanghai
  - Research Site, Shangqiu
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Weifang
  - Research Site, Wenzhou
  - Research Site, Xi'an
  - Research Site, Xiangtan
  - Research Site, Yantai
  - Research Site, Zhengzhou
  - Research Site, Zunyi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
  AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles.
  When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment https://vivli.org/. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/